CLINICAL TRIAL: NCT03372525
Title: Selective High Frequency Oscillation Ventilation(HFOV) vs Conventional Mechanical Ventilation(CMV) for Neonates With Acute Respiratory Distress Syndrome (ARDS) and/or RDS : a Randomized Controlled Trial
Brief Title: Invasive Ventilation Strategies for Neonates With Acute Respiratory Distress Syndrome Syndrome (ARDS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, Principal Investigator, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MV for ARDS
Record Dates: First submitted 2017-12-09; First posted 2017-12-13 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Acute Respiratory Distress Syndrome; Bronchopulmonary Dysplasia; High Frequency Oscillation Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: When the neonate had fulfilled the included criteria, selective HFOV or CMV were started immediately on the basis of the group assignment.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFOV (Experimental): Ventilated infants were randomized to HFOV.
  Interventions: Device: HFOV
- CMV (Active Comparator): Ventilated infants were randomized to CMV.
  Interventions: Device: CMV

INTERVENTIONS:
Device: HFOV — Infants were randomized to HFOV
  Arms: HFOV
Device: CMV — Infants were randomized to CMV
  Arms: CMV

SUMMARY:
Acute respiratory distress syndrome (ARDS) in neonates has been defined in 2017.The death rate is over 50%. HFOV and CMV are two main invasive ventilation strategies. However, which one is better needing to be further elucidated.

DETAILED DESCRIPTION:
Severe acute respiratory distress syndrome (ARDS) is one of the serious complications in critically ill neonates. It can result in severe hypoxemia refractory to mechanical ventilation. Usually, invasive ventilation with low parameters is enough for neonates with mild and moderate ARDS. And extracorporeal membrane oxygenation is used to neonates with severe ARDS. However, extracorporeal membrane oxygenation can also lead to high death rate and need more technique and conditions. Mechanical ventilation with higher parameters was a substitute for such situations, but the death rate, complications and injuries of higher parameters is unknown. The purpose of the present study was to compare HFOV with CMV as invasive respiratory support strategies on decrease the mortality and morbidities in neonate with ARDS.

ELIGIBILITY:
Inclusion Criteria:

* For a neonate to be included, the following four criteria must be fulfilled: (1)gestational age (GA) between 26+0 and 32+0 weeks (estimated on the postmenstrual date and early gestation ultrasonographic findings); (2)Birth weight less than 2000g; (3) assisted with CMV within 12 h after birth; (4)diagnosis with ARDS and/or RDS. (5)stabilization before randomization within 12 h after birth: FiO2<=0.30, pH>7.20, PaCO2<=60 mmHg, Paw <=7-8 cmH2O;

Exclusion Criteria:

* neonates with at least one of the following criteria are not eligible for the study: (1) Neonates who only needed noninvasive ventilation; (2) major congenital anomalies or chromosomal abnormalities; (3) neuromuscular diseases; (4) upper respiratory tract abnormalities; (5) need for surgery known before the first extubation; (6) Grade Ⅲ-IV-intraventricular hemorrhage (IVH); (7) congenital lung diseases or malformations or pulmonary hypoplasia.

Ages: 1 Minute to 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
bronchopulmonary dysplasia (BPD) | 28 days after birth or 36 weeks'gestational age or before discharge
  neonate was diagnosed with BPD
death | 28 days after birth or 36 weeks'gestational age or before discharge
  the included preterm infants were dead

SECONDARY OUTCOMES:
air leak | 28 days after birth or 36 weeks'gestational age or before discharge
  the included preterm infants were diagnosed with air leak
the incidence of retinopathy of prematurity(ROP) | 28 days after birth or 36 weeks'gestational age or before discharge
  the included preterm infants were diagnosed with ROP
the incidence of neonatal necrotizing enterocolitis(NEC) | 28 days after birth or 36 weeks'gestational age or before discharge
  the included preterm infants were diagnosed with NEC

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided